CLINICAL TRIAL: NCT04347837
Title: Multisite Study of Titan SGS Stapler in Longitudinal Gastric Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Standard Bariatrics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-2019-01
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Investigational device (Experimental): The investigational device will be used for all participants
  Interventions: Device: Titan SGS stapler

INTERVENTIONS:
Device: Titan SGS stapler — Stapler for the longitudinal resection of the stomach

SUMMARY:
The Titan SGS stapler is the first minimally invasive stapler designed for the longitudinal resection of the stomach. This is the first experience using this stapler in humans. The purpose of this study is to demonstrate use of the Titan SGS stapler in creating longitudinal gastric resection. Safety is defined by the absence of device related adverse events in the study period. Usability is evaluated based on surgeon evaluation of the device following each use.

This is a open label clinical trial to be conducted at three US sites. Up to 60 participants will be enrolled and will be followed for 6 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 to 65 undergoing a procedure requiring longitudinal gastric resection including: laparoscopic sleeve gastrectomy, laparoscopic gastric wedge resection, laparoscopic duodenal switch/loop duodenal switch.

Exclusion Criteria:

1. Age < 18 years
2. Incarceration
3. Prior gastric or foregut surgery (hiatal hernia repair, lap band +/- removal, Nissen fundoplication, gastrostomy tube, greater curve plication, sleeve gastrectomy etc.)
4. Diagnosed bleeding disorder (hyper or hypocoagulable state)
5. Systemic anticoagulation
6. Significant organ system disease

   1. Stage III CKD or greater
   2. Liver cirrhosis (any)
   3. CHG with EF < 50%
   4. COPD with O2 dependence
   5. Uncontrolled diabetes mellitus (A1C > 10%)
7. Intraoperative surgeon evaluation indicates the subject is not a candidate for longitudinal gastric resection with the Titan Stapler due to anatomic factors such as extensive abdominal adhesions or the device will not fit for the particular application.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Safety of the Titan SGS stapler | 6 weeks
  • Safety will be defined using descriptive statistics for device related adverse events in the study period.
Usability | 1 day
  • Usability of the Titan SGS to resect the stomach will be determined by the intraoperative assessment of the surgeon. The surgeon will complete a questionnaire with assessments of the device.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Kaleida Health Buffalo General Hospital, Buffalo, New York
  - WakeMed Bariatric Specialists of North Carolina, Cary, North Carolina
  - West Chester Hospital, West Chester, Ohio